CLINICAL TRIAL: NCT01734980
Title: Comparison Of Cytologic Accuracy Of Endobronchial Ultrasound Transbronchial Needle Aspiration Using Needle Suction Versus No Suction
Brief Title: Endobronchial Ultrasound Transbronchial Needle Aspiration Using Needle Suction Versus No Suction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Michel Chalhoub, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-018
Record Dates: First submitted 2012-07-04; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Mediastinal Lymphadenopathy; Lung Malignancies
Keywords: Endobronchial Ultrasound; transbronchial needle aspiration
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endobronchial Ultrasound (Experimental): EBUS-TBNA is a procedure that allows accurate sampling of mediastinal lymph nodes and peribronchial lesions
  Interventions: Procedure: Endobronchial Ultrasound

INTERVENTIONS:
Procedure: Endobronchial Ultrasound — The samples will be divided as 2 groups for comparison. Group A is the group of samples where we apply negative pressure syringe for needle suction. Group B is where no suction will be applied after needle insertion.

SUMMARY:
Cytological diagnostic accuracy between endobronchial ultrasonography endobronchial ultrasound transbronchial needle aspiration (EBUS-TBNA) samples using suction versus samples when no suction is applied.

DETAILED DESCRIPTION:
Endobronchial ultrasound-guided transbronchial needle aspiration which is known as the EBUS procedure is a low risk procedure performed using bronchoscopy to sample chest lesions. A needle is passed through the bronchoscope to biopsy the chest lesion. Every lesion is usually biopsied 3 to 7 times. In most cases the investigators apply a syringe with negative pressure to the needle inserted into lesion for biopsy. In some cases the investigators don't apply any negative pressure. There are no studies to evaluate which one is better, applying syringe suction or no suction.

In our study, the investigators are planning to do biopsies with or without suction. Then, the pathology samples will be evaluated for any cytologic difference in making the diagnosis. Any patient undergoing the EBUS procedure for chest biopsies will be eligible. Every lesion will be biopsied at least twice with needle with and without suction. The biopsy samples will be then divided into group A where the investigators applied syringe suction and group B where no syringe suction was applied. There is no risk to the patient in addition to the risk of the EBUS procedure itself. The investigators are not performing any additional intervention from the usual standard of care for any patient presenting for the EBUS procedure. Essentially the investigators are simply grouping the suction and no suction pathology samples as A and B for pathologic comparison.

RESULTS: Among the 26 participants, one of the patients (3.8%) had no adequate tissue using both methods; one patient (3.8%) had adequate tissue using suction but no adequate tissue using no suction; and 24 patients had adequate tissue using both methods (92.3%, p= 1.00). Among the twenty-four patients with adequate tissue using both methods, 14 patients (58.3%) had benign pathology using both methods, while ten patients (41.7%) had malignant pathology using both methods (p= 1.00). Considering suction to be the golden method, the sensitivity and specificity of no suction were 100%. Among the 32 sites that were sampled, one site (3.1%) had no adequate tissue using both methods; one site (3.1%) had adequate tissue using suction but no adequate tissue using no suction; and 30 sites had adequate tissue using both methods (93.8%, p= 1.00). Among the thirty sites with adequate tissue using both methods, 17 (56.7%) had benign pathology using both methods; 12 (40.0%) had malignant pathology using both methods; and one site (3.3%) had malignant pathology using suction, but benign pathology using no suction (p= 1.00). Considering suction to be the golden method, the no suction had a sensitivity= 92.3% and specificity= 100%.

ELIGIBILITY:
Inclusion Criteria:

* All adult subjects who are scheduled to undergo endobronchial ultrasound transbronchial aspiration to sample mediastinal masses or lymph nodes.

Exclusion Criteria:

* Patients who are not able to complete the EBUS procedure for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 3 days
  The number of patients with cytological diagnosis as a measure of effective diagnostic technique.

SECONDARY OUTCOMES:
Samples adequacy | 3 days
  adequate cytological material as a measure of effective diagnostic technique.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chalhoub, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States